CLINICAL TRIAL: NCT06573567
Title: Target Weight Guided by Bioimpedance Analysis in Hemodialysis Patients
Brief Title: Bioimpedance Analysis for Hemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cishan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, Han-ming Kuo, Director, Division of Nephrology, Cishan Hospital, Ministry of Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bioimpedance_hemodialysis
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioimpedance (Experimental): Use overhydration value obtained by bioimpedance analysis to guide fluid management; the measurements will be obtained once per month
  Interventions: Device: Bioimpedance
- Control (Placebo Comparator): Bioimpedance analysis done, but the results will be masked to the participants, care providers and outcome evaluators
  Interventions: Device: Control

INTERVENTIONS:
Device: Bioimpedance — Experimental: use overhydration value obtained by bioimpedance analysis to guide fluid management; the measurements will be obtained once per month
  Arms: Bioimpedance
Device: Control — Placebo Comparator: the measurements will also be obtained once per month, but not revealed to the participants and the care providers
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if bioimpedance-guided fluid management can help decrease hemodialysis complications. The main questions it aims to answer are:

Does bioimpedance-guided fluid management decrease major cardiovascular events? Does bioimpedance-guided fluid management decrease other hemodialysis complications?

Participants will:

Take bioimpedance analysis once per month Adjust dry weight according to the analysis as possible in active group Blind the analysis results to the doctor and the patient in the control group

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if bioimpedance-guided fluid management can decrease major adverse cardiovascular events (MACE), symptoms during hemodialysis, or other important outcomes such as vascular access patency, fluid overload admissions, etc. in maintenance hemodialysis patients. The main questions it aims to answer are:

Hypothesis 1: bioimpedance-guided fluid management decreases MACE Hypothesis 2: bioimpedance-guided fluid management decreases intradialytic hypotension, cramps and fatigue Hypothesis 3: bioimpedance-guided fluid management decreases need for urgent revascularization of vascular access for hemodialysis

Participants in the control group will decide their target weight according to physician's suggestion and the patient's preference, according to symptoms that are thought related to fluid status aberrancy (for example, edema, crackles for fluid overload, and cramps, intradialytic hypotension, fatigue for fluid insufficiency, given no other acute illness accountable for the symptoms and intradialytic weight gain not exceeding 5% of previous weight)

Participants in the active (bioimpedance) group will adjust their dry weight as those in the control group, if symptoms of fluid status aberrancy present. However, if no symptoms occur, they will receive adjustment according to measurements by bioimpedance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Has received hemodialysis >= 3 months
* Has at least 1 pair of intact same-side upper extremity and lower extremity

Exclusion Criteria:

* Pregnant
* With a cardiac pacemaker
* With metallic implants that may interfere with measurements (cardiac stents acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | From first bioimpedance analysis done to 1 year later
  A composite of myocardial infarction, stroke and all-cause mortality

SECONDARY OUTCOMES:
The number of hemodialysis sessions with intradialytic hypotension | From first bioimpedance analysis done to 1 year later
  During hemodialysis, systolic blood pressures (SBP) drop to <90mmHg, excluding those with baseline SBP <90mmHg
The number of hemodialysis sessions with intradialytic cramps or postdialytic cramps | From first bioimpedance analysis done to 1 year later
  Cramps during hemodialysis or later in the hemodialysis day, excluding those who experience cramps on non-hemodialysis day; cramps in both extremities and abdomen are counted
The number of hemodialysis sessions with pitting edema | From first bioimpedance analysis done to 1 year later
  Pitting edema is defined as grade 1 or more
The number of hemodialysis sessions with lung edema | From first bioimpedance analysis done to 1 year later
  Lung edema is defined as either of the followings:
  1. Crackles in lungs, excluding those with overt history or signs of other diseases that cause crackles, such as pneumonia, atelectasis or pleural disease
  2. Perihilar or interstitial pattern of infiltrations on chest X ray
The number of hemodialysis sessions with non-function of arteriovenous shunt | From first bioimpedance analysis done to 1 year later
  Non-function means absence of thrill or bruit of the shunt, and/or needle could not be placed with adequate blood flow for dialysis; both arteriovenous fistula and graft are considered in this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Han-Ming Kuo, Master, Study Chair — Cishan Hospital, MOHW, Taiwan
Locations (1):
- Cishan Hospital, MOHW, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.
Supporting Information: Study Protocol, SAP
Time Frame: one year after the research published
Access Criteria: The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Background] Liu L, Sun Y, Chen Y, Xu J, Yuan P, Shen Y, Lin S, Sun W, Ma Y, Ren J, Liu W, Lei J, Zuo L. The effect of BCM guided dry weight assessment on short-term survival in Chinese hemodialysis patients : Primary results of a randomized trial - BOdy COmposition MOnitor (BOCOMO) study. BMC Nephrol. 2020 Apr 15;21(1):135. doi: 10.1186/s12882-020-01793-x. PMID 32295531
- [Background] Onofriescu M, Mardare NG, Segall L, Voroneanu L, Cusai C, Hogas S, Ardeleanu S, Nistor I, Prisada OV, Sascau R, Covic A. Randomized trial of bioelectrical impedance analysis versus clinical criteria for guiding ultrafiltration in hemodialysis patients: effects on blood pressure, hydration status, and arterial stiffness. Int Urol Nephrol. 2012 Apr;44(2):583-91. doi: 10.1007/s11255-011-0022-y. Epub 2011 Jun 19. PMID 21688195
- [Background] Hur E, Usta M, Toz H, Asci G, Wabel P, Kahvecioglu S, Kayikcioglu M, Demirci MS, Ozkahya M, Duman S, Ok E. Effect of fluid management guided by bioimpedance spectroscopy on cardiovascular parameters in hemodialysis patients: a randomized controlled trial. Am J Kidney Dis. 2013 Jun;61(6):957-65. doi: 10.1053/j.ajkd.2012.12.017. Epub 2013 Feb 15. PMID 23415416
- [Background] Onofriescu M, Hogas S, Voroneanu L, Apetrii M, Nistor I, Kanbay M, Covic AC. Bioimpedance-guided fluid management in maintenance hemodialysis: a pilot randomized controlled trial. Am J Kidney Dis. 2014 Jul;64(1):111-8. doi: 10.1053/j.ajkd.2014.01.420. Epub 2014 Feb 28. PMID 24583055
- [Background] Huan-Sheng C, Yeong-Chang C, Ming-Hsing H, Fan-Lieh T, Chu-Cheng L, Tsai-Kun W, Hung-Ping C, Sze-Hung H, Hsien-Chang C, Chia-Chen L, Chun-Cheng H, Chun-Ting C, Hung-Hsiang L, Chun-Ju L, Paik-Seong L. Application of bioimpedance spectroscopy in Asian dialysis patients (ABISAD-III): a randomized controlled trial for clinical outcomes. Int Urol Nephrol. 2016 Nov;48(11):1897-1909. doi: 10.1007/s11255-016-1415-8. Epub 2016 Sep 12. PMID 27620902
- [Background] Patel HV, Annigeri RA, Kowdle PC, Rao BS, Seshadri R, Balasubramanian S, Vadamalai V. Bioimpedance Spectroscopy-Guided Ultrafiltration Normalizes Hydration and Reduces Intradialytic Adverse Events in Hemodialysis Patients. Indian J Nephrol. 2019 Jan-Feb;29(1):1-7. doi: 10.4103/ijn.IJN_150_18. PMID 30814786